CLINICAL TRIAL: NCT02370199
Title: Peripheral Blood Flow Responses to Electromagnetic Energy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nicole Lohr, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22652
Record Dates: First submitted 2015-02-18; First posted 2015-02-24 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Exposure to Man-made Visible Light
MeSH Terms: interventions — Ultraviolet Therapy; perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 670 nm light (Experimental): Subjects will have baseline blood flow measured in the gastrocnemius using octafluoropropane infusion and ultrasound.After baseline flow measurements are obtained, a 670 nm light emitting diode will be placed 1 cm above the gastrocnemius muscle. The diode will not be in direct contact with the skin. Subjects will be exposed to 75 mW/cm2. Contrast images will be obtained up to 5 minutes after the commencement of light.
  Interventions: Device: 670 nm light; Drug: octafluropropane

INTERVENTIONS:
Device: 670 nm light — 670 nm light emitting diode will be placed 1 cm above the gastrocnemius muscle. The diode will not be in direct contact with the skin. Subjects will be exposed to 75 mW/cm2.
  Other Names: Red light
Drug: octafluropropane — Octofluoropropane will be administered as a continuous infusion prior to the initiation of 670 nm light in order to measure skeletal muscle blood flow.
  Other Names: Definity

SUMMARY:
This study evaluates 670 nm energy in the form of red light to stimulate blood flow changes in healthy adults. All participants will receive red light to their leg. They will also receive a continuous infusion of Definity (octafluoropropane) ultrasound contrast.

DETAILED DESCRIPTION:
670 nm energy in the form of red light dilates isolated blood vessels. This study seeks to measure vessel dilation in human subjects exposed to this energy at different irradiance intensities (25 milliwatts (mW)/cm2 and 75 mW/cm2). The intent of this protocol is to measure blood flow in the gastrocnemius muscle before and after exposure to 670 nm light energy. This protocol will be performed in healthy subjects, who do not meet exclusion criteria. The study consists of one visit. Blood flow measurement will be performed using contrast enhanced ultrasound, a method by which ultrasound contrast is continuously infused into the blood stream. Ultrasound records images in the area of interest and flow is related to the intensity of the contrast in each image. After baseline blood flow images are collected, the subject will receive red light energy to the gastrocnemius muscle with concurrent blood flow measurements with contrast ultrasound. The subject will be monitored post procedure and the study will then be completed.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be healthy subjects over the age of 18.
* Men and women will be recruited for participation.
* All ethnicities will be included in this study.

Exclusion Criteria:

Exclusionary criteria include:

* age under 18 years and those over 60 years of age,
* those who are unable to understand the consent process,
* those who cannot read or speak English,
* a history of cancer,
* peripheral artery disease,
* diabetes mellitus,
* active pregnancy,
* hypersensitivity to perflutren contrast agents,
* pulmonary hypertension,
* chronic kidney disease,
* active tobacco or drug use,
* blood pressure over 160/90, BMI>30,
* sickle cell disease, or
* history of intracardiac shunt.

Additional exclusion criteria include:

* a history of coronary artery disease,
* heart failure,
* the presence of an implanted defibrillator or pacemaker,
* a history of heart murmur or rhythm disorder (atrial fibrillation, atrial tachycardia, or ventricular tachycardia),
* neurological diseases such as stroke, and
* any uncontrolled medical conditions.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in blood flow (using octafluoropropane infusion and ultrasound) | 10 minutes
  Blood flow changes based on ultrasound imaging

CONTACTS AND LOCATIONS:
Overall Officials: Nicole L Lohr, MD, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States